CLINICAL TRIAL: NCT05470166
Title: Lidocaine Infusion With Enhanced Recovery Program for Pancreatic Cancer Surgery: Effect on Pain and Patient Immunity
Brief Title: Lidocaine Infusion With ERAS Protocol for Pancreatic Cancer Surgery: Effect on Pain and Patient Immunity.
Acronym: ERAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: University of Alexandria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: lidocaine ERAS whipple
Record Dates: First submitted 2022-06-02; First posted 2022-07-22 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2022-04

CONDITIONS: ERAS; Lidocaine; Cancer of Pancreas; Natural Killer Cell Cytokine Production
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- infusion of intraoperative lidocaine to patients undergoing whipple surgery (Experimental): lidocaine 1.5mg/kg infused as bolus, then 2mg/kg/hr through the operation
  Interventions: Drug: Lidocaine IV
- saline infusion of same volume of lidocaine (Experimental): same amount of normal saline infused as bolus and infusion
  Interventions: Other: saline IV

INTERVENTIONS:
Drug: Lidocaine IV — lidocaine infusion as bolus 1.5mg/kg then 2mg/kg/hr
  Arms: infusion of intraoperative lidocaine to patients undergoing whipple surgery
Other: saline IV — saline infusion same volume as lidocaine
  Arms: saline infusion of same volume of lidocaine

SUMMARY:
The whole world now is directed to implement strategies that enhance the patient's quality of life and prevent tumor relapse.

Enhanced recovery after pancreatic surgery (ERAPS) program was found to improve the quality of life as it is an evidence-based protocol designed to standardize and optimize perioperative medical care in order to reduce surgical trauma, perioperative physiological stress, organ dysfunction, reduction of clinical complications, length of hospital stay and the health costs together with increase of patient satisfaction.

lidocaine; it is an amide local anaesthetic Recently its use as intravenous perioperative infusion for abdominal cancer surgeries is encouraging, as it significantly reduces postoperative pain, opioid consumption and nausea and vomiting. it also promotes gastrointestinal function recovery, and shortens the postoperative hospital stay. In addition, lidocaine in particular can act directly and indirectly on pancreatic cancer cells and the tumor microenvironment.

The investigators suggest that IV lidocaine infusion in combination with ERAPS protocol may achieve better postoperative outcomes after pancreatic surgery for cancer.

DETAILED DESCRIPTION:
The whole world now is directed to implement strategies that enhance the patient's quality of life and prevent tumor relapse , so the Enhanced recovery after pancreatic surgery (ERAPS) program was found to improve the quality of life as it is an evidence-based protocol designed to standardize and optimize perioperative medical care in order to reduce surgical trauma, perioperative physiological stress, organ dysfunction, reduction of clinical complications, length of hospital stay and the health costs together with increase of patient satisfaction.

ERAPS was applied for pancreatic surgery in 2012, since that time 27 developed ERAPS items were evaluated, 5 of them got the highest level of evidence those include (avoiding hypothermia, use of wound catheters for continuous analgesia, antimicrobial, thromboprophylaxis protocols and preoperative nutritional interventions for patients with severe weight loss (15%). ERAS society encourages further researches to improve compliance and outcome and to confirm the benefit of current updated recommendations.

Many drugs had been used in the anaesthetic management of major abdominal surgeries and of which is lidocaine; it is an amide local anaesthetic commonly used for regional and neuraxial blocks. Recently its use as intravenous perioperative infusion for abdominal cancer surgeries is encouraging, as it significantly reduces postoperative pain, opioid consumption and nausea and vomiting. it also promotes gastrointestinal function recovery, and shortens the postoperative hospital stay.

In addition, lidocaine in particular can act directly and indirectly on pancreatic cancer cells and the tumor microenvironment. At the tumor level, lidocaine can induce apoptosis in cancer cells by inhibiting Src phosphorylation and reducing the expression of adhesion molecules. In the tumor microenvironment, lidocaine can enhance the activity of immune cells such as natural killer cells, which are responsible for directly attacking cancer cells. Furthermore the impact of lidocaine on post-operative opioid consumption could be another factor that reduces the opioid associated cancer progression.

Natural killer (NK) cells are cluster of differentiation 3 (CD3-) -cluster of differentiation 56 (CD56+) lymphocytes playing a pivotal role in the innate immune response against cancer. Their main purpose is identification and eradication of virus infected cells and metastatic cells. Diminished activity of NK cells is a predisposing factor for cancer recurrence. Preservation of innate immune function and the direct anti-inflammatory effects may be the cause of the protective effects of local anaesthetics and regional techniques.

Different concentrations of local anaesthetics appear to have different effects on NK cytotoxicity. High concentrations of lidocaine suppress NK cell cytotoxicity; yet clinically relevant concentrations enhance the in vitro function of NK cells via the release of lytic granules. Hence, lidocaine appears to have predominantly anticancer effects So the investigators suggest that IV lidocaine infusion in combination with ERAPS protocol may achieve better postoperative outcomes after pancreatic surgery for cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-70 years
2. Both sex.
3. American society of anesthesiology (ASA) physical status class II;III.
4. Resectable pancreatic tumors.

Exclusion Criteria:

1. Patients with history of sensitivity to lidocaine,
2. Diabetic patients.
3. Body weight loss > 15%.
4. Opioid tolerant patient or patient receiving nonsteroidal anti-inflammatory drugs within 1 week of surgery or antiarrythmic drugs.
5. Cognitive dysfunction.
6. Any history of antitumor treatments or chemotherapy before surgery
7. Any contraindication for neuraxial anaesthesia.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Post-operative nociceptive pain assessment. | 24 hours postoperative
  post operative pain assessment using visual analogue scale (VAS), The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be.

SECONDARY OUTCOMES:
Effect on immune response | pre-operative and 5 days postoperative
  Natural killer cell isolation will be done preoperatively and 5 days postoperative
Effect on i tumor recurrence | pre-operative and 5 days postoperative
  cytotoxic lymphocytes assay will be measured preoperatively and 5 days postoperative
Total intra-operative fluid requirements. | intra-operative every 10 minutes
  Total intraoperative fluid requirements in liters and fluid responsiveness assessed by pleth variability index (PVI) every 10 minutes to keep value < 13 %.
Gastro-intestinal recovery. | up to 5 days postoperative
  effect of lidocaine on enhancing gastrointestinal motility,Time to return of bowel sounds in hours, first time to pass flatus and time to first defecation in hours will be recorded.
Time to first ambulation | up to 5 days post-operative
  effect of lidocaine and epidural analgesia on pain
Total analgesic consumption | up to 5 days post-operative
  effect of lidocaine on analgesic requirements
Length of hospital stay in days | up to 5 days postoperative
  effect of lidocaine on ERAS and Duration of hospital stay in days will be recorded in both groups including the start of the hospitalization time
Effect on haemodynamics | intraoperative and 5 days post-operative
  effect of lidocaine on heart rate in beats per minute
Effect on haemodynamics | intraoperative and 5 days post-operative
  effect of lidocaine on blood pressure in mmHg
Perioperative complications | intraoperative and up to 5 days postoperative
  recording of any complications perioperatively and postoperatively Nausea and vomiting, wound infection, urinary tract infection, deep vein thrombosis and hematoma will be recorded in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
through clinical trials
Supporting Information: Study Protocol, SAP
Time Frame: 6 months up to 1 year
Access Criteria: Lidocaine ERAS whipple surgery patient immunity